CLINICAL TRIAL: NCT02179840
Title: Assessment of Coherent Hemodynamics Spectroscopy (CHS) as a New Tool for Monitoring Cerebral Blood Flow and Autoregulation at the Microvascular Level
Brief Title: Assessment of Cerebral Microvascular Circulation
Acronym: CHS-Brain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not initiated, no participants enrolled.
Sponsor: University of California, San Francisco (Other)
Collaborators: Tufts University (Other); University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHS-Brain
Record Dates: First submitted 2014-06-23; First posted 2014-07-02 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Cerebral Microvascular Circulation
Keywords: Cerebral microvascular circulation; Cerebral autoregulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous (Active Comparator): Anesthesia is maintained via intravenous agents. Mechanical ventilation adjustment will be performed.
  Interventions: Procedure: Mechanical ventilation adjustment
- Inhalational (Active Comparator): Anesthesia is maintained via inhalational agents. Mechanical ventilation adjustment will be performed.
  Interventions: Procedure: Mechanical ventilation adjustment

INTERVENTIONS:
Procedure: Mechanical ventilation adjustment — Mechanical ventilation adjustment and study procedure: This is a validation study of the CHS method in assessing cerebral microvascular hemodynamic changes. Cyclical physiological events such as respiration are essential in CHS methodology. The previous study shows that the robust measurement of the CHS method occurs at a respiratory rate of about 4-10 breaths per minute. Therefore, we propose the following respiration adjustment in this study with the consideration that CO2 is a powerful regulator of cerebral blood flow. Blood gas analysis will be performed during the 1st and 2nd rounds of ventilation adjustment.

SUMMARY:
One of the fundamental goals of anesthesia care is to optimize tissue perfusion and oxygenation, especially in critically ill patients. The standard monitors such as blood pressure, heart rate and pulse oximetry do not directly reflect tissue information and can be misleading sometimes. Coherent hemodynamics spectroscopy (CHS) based on cerebral oximetry is proposed as a continuous and non-invasive tool assessing cerebral microvascular hemodynamics. The investigators propose this study to explore the validity of CHS via comparison with transcranial Doppler measurement in anesthetized surgical patients. The hypotheses are: 1) CHS can effectively measure cerebral microvascular hemodynamic changes associated with mechanical ventilation adjustment during anesthesia. 2) CHS can assess functional status of cerebral autoregulation that is altered by hypercapnia and inhalational anesthetic agent.

DETAILED DESCRIPTION:
One of the essential goals in taking care of anesthetized surgical patients is to maintain adequate tissue perfusion and oxygenation. This is especially true for vital organs like the brain. Unfortunately, neither cerebral oxygen consumption nor cerebral oxygen delivery are directly monitored in the clinical setting while this type of information is of particular importance when taking care of patients inflicted with critical neurologic conditions. In addition, cerebral autoregulation - the mechanism of maintaining a constant cerebral blood flow in the face of arterial blood pressure fluctuation, is also not routinely monitored. The recent establishment of Coherent Hemodynamics Spectroscopy (CHS) is promising in offering what is needed in this context. The uniqueness of CHS is that it does not add any additional monitoring modality other than the cerebral oximeter based on near-infrared spectroscopy (NIRS) that is currently used in clinical care. However, CHS is based on its own innovative algorithm that quantifies microvascular cerebral blood flow and oxygen consumption, separates arterial and venous blood, and assesses functional status of cerebral autoregulation while the conventional cerebral oximeters do not. The investigators have established collaborations with Dr. Fantini from Tufts University and Dr. Tromberg from Beckman Laser Institute who are both leading scientists in Biophotonics research and development. Based on the clinical strength at UCSF, it is the investigators collaborative plan to explore the clinical application of CHS in patients with and without intracranial pathophysiologies. The study protocol has been submitted for review at UCSF.

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18 years of age or older
* Relative healthy (ASA I-II)
* Scheduled for elective intra-abdominal surgeries including colorectal, urological and gynecological procedures under general anesthesia with placements of endotracheal tube and radial arterial catheter.
* Paralysis is required for surgery
* A total of 30 patients will be recruited. These 30 patients are randomly divided into 2 groups based on the technique of anesthesia maintenance during surgery. The anesthesia in one group (n=15) is maintained using inhalational agent. The anesthesia in the other group (n=15) is maintained using intravenous agents.

Exclusion Criteria:

* Patients <18 years of age
* ASA physical status ≥III
* Emergent or urgent surgery
* Laparoscopic surgery
* History of pulmonary diseases including COPD
* Asthma
* Restrictive lung disease, etc.
* History of cardiac diseases including symptomatic coronary artery disease, heart failure, arrhythmia, moderate to severe valvular abnormalities, and cardiomyopathies
* History of neurological diseases including carotid artery disease, stroke or TIA, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
cerebral oximetry | 3 minutes following the intervention
  Cerebral blood flow capillary transit time and cerebral autoregulation

CONTACTS AND LOCATIONS:
Overall Officials: Lingzhong Meng, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States